CLINICAL TRIAL: NCT01328340
Title: The Effect of High-speed Power Training on Muscle Performance, Function and Pain in Older Adults With Knee OA
Brief Title: High-speed Power Training in Older Adults With Knee Osteoarthritis (OA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Collaborators: American College of Rheumatology (Other); Arthritis Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 1043138
Record Dates: First submitted 2011-03-31; First posted 2011-04-04 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-10

CONDITIONS: Knee Osteoarthritis
Keywords: muscle power, exercise, aging
MeSH Terms: conditions — Osteoarthritis, Knee; Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- High-speed power training (Active Comparator): Volunteers randomized into SHPT will be exercised 3 times per week for 12 weeks. Each training session will consist of 3 sets of 12 to 14 repetitions at 40% of maximal strength for leg press (LP) and seated knee extension (KE) exercises.
  Interventions: Other: High-speed power training
- Slow-speed strength training (Active Comparator): Volunteers randomized into STR will be exercised 3 times per week for 12 weeks. Each training session will consist of 3 sets of 8 to 10 repetitions at 80% of maximal strength for LP and KE exercises.
  Interventions: Other: Slow-speed strength training
- Control (No Intervention): Volunteers randomized into CON will undergo a placebo exercise intervention consisting of lower extremity range of motion and flexibility exercises performed 2 times per week with the assistance of the research staff.

INTERVENTIONS:
Other: High-speed power training — exercised 3 times per week for 12 weeks. Each training session will consist of 3 sets of 12 to 14 repetitions at 40% of maximal strength
  Other Names: weight training
  Arms: High-speed power training
Other: Slow-speed strength training — exercised 3 times per week for 12 weeks. Each training session will consist of 3 sets of 8 to 10 repetitions at 80% of maximal strength
  Other Names: weight training
  Arms: Slow-speed strength training

SUMMARY:
We are exploring a unique weight-training program for men and women 55 years or older with knee osteoarthritis (OA) that emphasizes high-speed movements. We believe that the speed at which muscles move may be more important to the improvement of muscle performance, function and pain than how strong the muscles are. We are comparing high-speed power training with traditional strength training to determine which method has the greatest effects on muscle strength, muscle power, speed of movement, functional performance and pain. We believe that high-speed training will improve these measures to a greater extent than simply training for increased muscle strength.

DETAILED DESCRIPTION:
The study compared 12 weeks of explosive high-speed power training with traditional slow-speed strength training. Outcome measures included muscle performance: leg press (LP) and knee extension (KE) one-repetition maximum (1RM) and LP peak power (PP), velocity at peak power (PPV) and force at peak power (PPF) from 40%-90% of the 1RM. Measures of function consisted of the 400-meter walk (400-m W), Berg Balance Scale (BBS), timed chair rise (TCR) and self-reported function and pain using the WOMAC.

Participants reported to the laboratory for 2 weeks of baseline measurements. On visit 1, subjects were explained the study and completed an informed consent document. On visit 2 and 3, muscle performance and functional measures were obtained. The following week, all muscle performance and functional measures were repeated to establish reliability. At the end of baseline testing, participants were randomized to treatment. Following the 12-week RT intervention, post-training muscle performance and functional measures were obtained.

Resistance Training Protocol. Volunteers randomized into high-speed power training (HSPT) and slow-speed strength training (SSST) exercised 3 times per week for 12 weeks using computer-interfaced Keiser a420 pneumatic leg press and knee extension RT equipment (Fresno, CA). For HSPT, each training session consisted of 3 sets of 12-14 repetitions at 40%1RM. Participants performed an explosive movement at high speed during the concentric phase of each repetition, paused for one-second, and performed the eccentric portion of the contraction over 2 seconds. Volunteers randomized into SSST also exercised 3 times per week for 12 weeks with each training session consisting of 3 sets of 8-10 repetitions at 80%1RM. The participants performed each movement at a slow velocity (2 s for concentric phase of the repetition), paused for one second, and performed the eccentric portion of the contraction over 2 seconds. CON met three times a week for warm-up and stretching exercises, but performed no RT. HSPT and SSST participated in the same warm-up and stretching exercises as CON.

Measures Maximal strength and power. Leg press and seated knee extension 1RM were obtained using Keiser pneumatic RT equipment fitted with a420 electronics. The seat of both the recumbent LP and KE apparatus was positioned to place the hip and knee joints between 90 and 100 degrees of flexion. The 1RM was obtained by progressively increasing resistance until the subject was no longer able to push out one repetition successfully. The Borg Scale was used to assist in evaluating when 1RM (combined with perceived maximal effort) was reached. Peak muscle power was obtained at 40%, 50%, 60%, 70%, 80% and 90% of the 1RM approximately 30 minutes after 1RM testing (8,9). Participants were instructed to exert "as fast as possible" at each relative percentage of the 1RM. Three attempts were made at each resistance and the greatest PP output obtained at each resistance was used in the analysis. The corresponding PPV and PPF were obtained for each external resistance from 40%-90% 1RM. The 1RM was measured bi-weekly in HSPT and SSST only and relative training intensity was adjusted accordingly to ensure adequate overload during training. Post-training muscle performance measures were obtained using loads relative to the initial baseline 1RM as well as the post-training 1RM.

400 meter self-paced walk (400-m W). Participants were instructed to walk at a pace they could maintain without overexerting themselves until they complete the 400-m W or could no longer continue. Standardized verbal encouragement was given at 30-second intervals during the walk. Participants taking longer than 15 minutes to complete the 400-m W were considered unable to successfully perform the test.

Berg Balance Scale (BBS). The BBS consists of 14 tests of balance scored on a 0-4 scale that are summed to obtain an aggregate balance score (range=0-56).

Timed Chair Rise (TCR). Volunteers placed their folded arms across their chests and stood up from a sitting position as an initial assessment. If subjects were able to accomplish this task, they were then asked to complete a timed bout of five repetitions with the instructions to complete the activity as fast as they can. Subjects completed the activity from the same armless chair (height of seat 43.18 cm). TCR was reported as the number of repetitions per minute calculated from the time required to complete five chair stands.

WOMAC Function and Pain. Self-reported function was assessed by the WOMAC function subscale, a 17-item Likert scale questionnaire (0=none, 1=mild, 2=moderate, 3=severe, 4=extreme) and pain was assessed by the WOMAC pain subscale, a 5-item Likert scale questionnaire (0=none, 1=mild, 2=moderate, 3=severe, 4=extreme). Self-reported function was represented by summation of the component item scores (range: 0-68; higher scores indicate greater functional loss) and pain was represented by summation of the component item scores (range: 0-20; higher scores indicating greater levels of pain).

ELIGIBILITY:
Inclusion Criteria:

* 55 years of age
* physician diagnosed knee OA
* relatively inactive
* male or female
* good overall health
* living independently (not in a nursing home or care facility)

Exclusion Criteria:

* heart attack or unstable angina within 6 months of consent
* hip fracture, knee or hip replacement within 6 months of consent
* diagnosed neurological disease
* pulmonary disease requiring use of oxygen
* osteoarthritis of the knee
* severe visual or hearing impairment

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2005-06; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Strength and power | 3 months
  The strength of the lower limb muscles will be measures using Keiser pneumatic leg press and knee extension exercise machines. The Keiser machines allow for the specific measurement of the contributions of force and velocity to the development of power, which will reveal whether the high-speed training protocol impacts speed-related measures of muscle performance.

SECONDARY OUTCOMES:
Function | 3 months
  Measures of mobility and function were evaluated using the 400-m Walk, Berg Balance Scale and timed chair rise which assess walking endurance, balance, and strength, respectively, all important variables for mobility

CONTACTS AND LOCATIONS:
Overall Officials: Stephen P Sayers, PhD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sayers SP, Gibson K, Cook CR. Effect of high-speed power training on muscle performance, function, and pain in older adults with knee osteoarthritis: a pilot investigation. Arthritis Care Res (Hoboken). 2012 Jan;64(1):46-53. doi: 10.1002/acr.20675. PMID 22012877